CLINICAL TRIAL: NCT02886364
Title: Evaluation of the Adapted Safe Childbirth Checklist and Respectful Care in Rural Community Hospitals and Maternity Centers in Chiapas, Mexico: A Mixed Methods Convergent Intervention Study
Brief Title: Adapted Safe Childbirth Checklist in Chiapas, Mexico
Acronym: SCC-Chiapas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Palazuelos, Associate Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P000000
Record Dates: First submitted 2016-08-28; First posted 2016-09-01 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy; Childbirth; Quality of Care; Puerperium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women delivered at AAC Hospital (Other): The intervention is only being implemented at the Ángel Albino Corzo Hospital due to limited funding. The site was selected by the Ministry of Health in Chiapas as a hospital that would benefit from improved quality of care around childbirth. There are no other arms in this study.
  Interventions: Behavioral: Adapted Safe Childbirth Checklist

INTERVENTIONS:
Behavioral: Adapted Safe Childbirth Checklist — The World Health Organization has created and endorsed the WHO Safe Childbirth Checklist as a tool for improving quality of care around childbirth. This tool has been modified to the context in Mexico by another group of investigators at the National Institute of Public Health. Our team expanded the Mexican version of the WHO Safe Childbirth Checklist to include indicators around respectful maternity care.

SUMMARY:
The purpose of this mixed methods study is to evaluate the implementation of an adapted Safe Childbirth Checklist in a rural hospital in Chiapas, Mexico. The study aims are:

1. To evaluate the implementation of the adapted Safe Childbirth Checklist using quality of care indicators and the perspectives of providers and patients;
2. To examine changes in the perceptions of disrespectful and respectful practices around childbirth among providers before and after a quality improvement program.
3. To understand how postpartum women and their male partners perceive the care they received at the hospitals in Ángel Albino Corzo and Revolución with regard to disrespectful and respectful practices, and how, if at all, these experiences compare with prior birth experiences in other settings.
4. To examine trends in proportion of facility-based births in the catchment area of the hospital after the implementation of the adapted Safe Childbirth Checklist

DETAILED DESCRIPTION:
This is a mixed methods convergent intervention study design. Quantitative and qualitative data will be collected and integrated to answer the specific aims above. There are 3 groups of people who will be approached to participate in this study:

1. Obstetric providers at the maternity center in Revolución (approximately 7-15 people)
2. Pregnant women who come to the maternity center or hospitals in Ángel Albino Corzo or Revolución to give birth from September 2016 - June 2017 (approximately 300 women, age >15 years old)
3. Postpartum women who delivered in the maternity center or hospitals after September 2016 (approximately 30-40 women, age >15 years old) and their male partners (approximately 30-40 men, age >15 years old) who live in Partners In Health-affiliated communities

The quality improvement training program will center on coaching around the adapted Safe Childbirth Checklist. This document contains reminders for evidence-based practices during childbirth, and it has been adapted to the context in Mexico. Only standard of care practices will be taught and employed at the maternity center. The quality improvement program has no additional intervention that would change diagnoses or management during peripartum care.

Risks to subjects are minimized by ensuring privacy in all research encounters. Additionally, research staff will not provide any clinical care to subjects, thereby dissociating participation in research from receiving clinical care.

There are no anticipated harms to the participants of this study that would compromise their safety because our quality improvement program does not introduce a new diagnostic test or treatment modality. The only foreseeable risk is emotional distress from discussing a potentially traumatic birth experience, which could occur with both healthcare providers and patients. The research team will undergo sensitization training in identifying signs of distress that may arise during the survey, interview, or focus group. They will be instructed to provide the appropriate mental health referrals if necessary. Partners In Health has a growing mental health program that can provide appropriate clinical accompaniment if required.

The investigators are restricting the study specifically to women who have an opportunity to benefit from the results of the study because they live in the catchment area of the maternity center and may seek childbirth care there in the future. The investigators are only including the providers at a single maternity center because that is the facility where Partners In Health has an affiliation and leads the quality improvement training program. Participants who do not stand to benefit from the results due to geographic or political barriers will not be included. All research will be conducted in Spanish. Non-Spanish speaking women are rare in this area, and will have to be excluded from the study due to the lack of trained interpreters in indigenous languages in the area.

Food will be provided at all focus groups. Postpartum women and their partners who consent to participate in interviews will receive a small token of appreciation, such as a bag of beans, bag of rice, or a bottle of cooking oil. These remunerations are thought to be appropriate for the cultural setting and are not large enough to be coercive.

All consents will be done by trained research staff, not by clinical staff, to avoid coercion. The obstetric providers will be asked to provide written consent, as they are literate. The postpartum women and their partners will provide verbal consent, as the majority are illiterate.

The adapted Safe Childbirth Checklist and discharge survey will be programmed into a mobile application on CommCare, which provides a secure cloud for data capture. Only research staff responsible for direct data analysis will have access to this secure data cloud.

The focus groups and interviews will be audio-recorded, transcribed in Spanish, and translated into English. All personally identifiable information will be removed. These files will be saved on an encrypted computer and only shared with research members through secure firewalls.

There will be one master file that lists the participants names and unique study ID number, so that responses can be linked longitudinally for providers and patients. Only the principal and lead investigators will have access to this file, which will be kept on an encrypted computer and deleted at the end of the study.

A Partners In Health team manager will provide ongoing supervision of the trained study staff and will be available to ensure appropriate data collection and trouble-shoot any questions or difficulties. The PI, funders, and site directors will review any adverse events to address potential areas of improvement.

No survey or focus group or interview transcript will contain personally identifiable information. The name of the participant and her community of residence will be kept in a secure Excel file linked to a unique study ID. The study ID will be used on all research related materials.

All data will be saved on encrypted computers, and files will only be shared behind a secure firewall. Only investigators who are directly involved in data collection and analysis will have access to these files.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivered at Ángel Albino Corzo Hospital between September 2016 and June 2017
* Women who live in Partners In Health-affiliated communities

Exclusion Criteria:

* Index pregnancy that ended in miscarriage or stillbirth
* Non-Spanish speaking

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Perceptions of patient safety and quality of care from providers and patients | 10 months
  Qualitative data will be collected through interviews of providers, postpartum women and their partners regarding their childbirth experiences in the district hospital where the adapted Safe Childbirth Checklist was implemented.
Adherence with evidence-based practices in the checklist | 10 months
  Quantitative data will be collected through key indicators in the checklist to capture uptake of best practices over time.
Number of facility-based childbirths within Partners In Health-affiliated communities in the catchment area of hospital | 10 months
  The proportions of facility-based births vs. home births will be compared pre- and post-implementation of the adapted Safe Childbirth Checklist.

IPD SHARING:
Plan to Share IPD: No